CLINICAL TRIAL: NCT00080470
Title: Battery Powered Bion Clinical Investigation: An Implantable Microstimulator for the Chronic Treatment of Refractory Urinary Urge Incontinence
Brief Title: An Implantable Microstimulator for the Chronic Treatment of Refractory Urinary Urge Incontinence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR-B-001
Record Dates: First submitted 2004-04-01; First posted 2004-04-05 (Estimated); Results first posted 2013-10-10 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-10

CONDITIONS: Urinary Incontinence
Keywords: Incontinence; Refractory; Urinary; Urge; Stimulation; Nerve; Microstimulator; Neuromodulation
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Stimulation On from Initial Activation up to the 12 month post-activation. Stimulation Off from 12 months post-activation until 45 days after the 12 month visit. Stimulation On from 45 days post 12 month visit and on.
  Interventions: Device: bion
- 2 (Sham Comparator): No Stimulation until 45 days post-implant. Stimulation On from 45 days post-implant and on.
  Interventions: Device: bion

INTERVENTIONS:
Device: bion — battery powered microstimulator

SUMMARY:
This clinical trial is being conducted to investigate the safety and effectiveness of a new device designed to treat urinary urge incontinence in those patients who have tried and failed two or more conservative therapies.

ELIGIBILITY:
Key Inclusion Criteria:

1. Age 18 years and above.
2. Diagnosed with urinary urge incontinence.
3. Have no reported history of urethral obstruction/stricture, bladder calculi or bladder tumor.
4. Have normal upper urinary tract function.
5. Be capable of giving informed consent.
6. Be capable and willing to follow all study related procedures.

Key Exclusion Criteria:

1. Have any active implantable device regardless of whether stimulation status is ON or OFF.
2. Are pregnant as confirmed by a urine pregnancy test or plan to become pregnant during the following 12 months period.
3. Less than one year post partum and/or are breast-feeding.
4. Have any passive implant that contains metal or electrically conductive materials.
5. Have conditions requiring Magnetic Resonance Imaging (MRI) evaluation.
6. Have conditions requiring diathermy procedures.
7. Have an inability to operate the bion Remote Control and bion Recharging System either by self or caregiver.
8. Have diabetes with peripheral nerve involvement or have severe uncontrolled diabetes.
9. Have history of coagulopathy or bleeding disorder.
10. Have a history of pelvic pain as primary diagnosis.
11. Have anatomical restrictions such that the study device placement is not possible.
12. Are currently participating or have participated within the past 30 days in any clinical investigation involving or impacting urinary or renal function.
13. Have a life expectancy of less than 1 year.
14. Cannot independently comprehend and complete the QoL questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2003-06; Primary Completion 2008-07 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Baynham, PhD, Study Director — Boston Scientific, Neuromodulation
Locations (11):
- United States (11):
  - Arizona Health Sciences Center (University of Arizona), Tucson, Arizona
  - The Department of Urology, Stanford University Medical Center, Stanford, California
  - Milestone Medical Research, Englewood, Colorado
  - Bladder Control Center of Norwalk, Norwalk, Connecticut
  - Walter Reed Army Medical Center, Division of Pelvic Medicine and Reconstructive Surgery, Washington D.C., District of Columbia
  - William Beaumont Hospital, Royal Oak, Michigan
  - Cornerstone Medical Specialty Center, Woodbury, Minnesota
  - The Pelvic and Sexual Health Institute (affiliated with Graduate Hospital), Philadelphia, Pennsylvania
  - Dallas Center for Pelvic Medicine, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Sound Urological Associates, Edmonds, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Although enrollment numbers totaled 148 subjects, the total number of implanted subjects were used for the analysis. Total number of implanted subjects is 87.
Groups:
- Treatment: Stimulation On from Initial Activation up to the 12 month post-activation. Stimulation Off from 12 months post-activation until 45 days after the 12 month visit.
  Stimulation On from 45 days post 12 month visit and on.
- Control: No Stimulation from post-implant until 45 days post-implant. Stimulation On from 45 days post-implant and on.
Period: Overall Study
Arm/Group | Treatment | Control
Started | 45 | 42
Completed | 11 | 14
Not Completed | 34 | 28

BASELINE CHARACTERISTICS:
Groups:
- Control: No stimulation until 45 days post-implant. Stimulation On from 45 days post-implant and on.
- Total: Total of all reporting groups
Arm/Group | Control | Treatment | Total
Number analyzed (Participants) | 42 | 45 | 87
Age, Customized [Mean (Standard Deviation); unit: Years] | 59.26 (12.66) | 54.82 (16.73) | 56.97 (14.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 40 | 81
  Male | 1 | 5 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Leaks Per Day
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Number of Leaks Per Day
Arm/Group | Treatment | Control
Number analyzed (Participants) | 45 | 42
Number of Leaks Per Day | NA (NA) — This study was limited by poor adherence to the clinical protocol and by incomplete data recovery. Data related to clinical effectiveness was not recoverable. Analysis of efficacy-related endpoints was not possible. | NA (NA) — This study was limited by poor adherence to the clinical protocol and by incomplete data recovery. Data related to clinical effectiveness was not recoverable. Analysis of efficacy-related endpoints was not possible.

2. Primary Outcome: Freedom From Major Complications
Time Frame: 5 years
Measure: Number; unit: Number of Adverse Events
Arm/Group | Treatment | Control
Number analyzed (Participants) | 45 | 42
Number of Adverse Events | 0 (NA) | 0 (NA)

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Control | Treatment
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/45
Other Adverse Events (participants affected / at risk) | 35/42 | 32/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=42) | Treatment (N=45)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal Discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 2 (3) | 0 (0)
Adhesion (General disorders) | 1 (1) | 0 (0)
Implant Site Pain (General disorders) | 2 (2) | 3 (3)
Implant Site Paresthesia (General disorders) | 0 (0) | 1 (1)
Therapeutic Product Ineffective (General disorders) | 17 (18) | 13 (16)
Therapeutic Response Decreased (General disorders) | 5 (5) | 4 (5)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 2 (2)
Vaginal Infection (Infections and infestations) | 1 (1) | 0 (0)
Device Breakage (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Device electrical Finding (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Device Failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Device Migration (Injury, poisoning and procedural complications) | 4 (4) | 2 (3)
Failure of Implant (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Inappropriate Device Stimulation of Tissue (Injury, poisoning and procedural complications) | 1 (1) | 6 (6)
Incision Site Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Suture Related Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle Spasm (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculuskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Dysaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Muscle Contractions involuntary (Nervous system disorders) | 3 (3) | 7 (8)
Nerve Compression (Nervous system disorders) | 1 (1) | 1 (1)
Neurological symptom (Nervous system disorders) | 1 (2) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urge Incontinence (Renal and urinary disorders) | 1 (1) | 3 (3)
Genital Pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic Discomfort (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic Pain (Reproductive system and breast disorders) | 3 (3) | 3 (3)
Perineal Pain (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Vaginal Pain (Reproductive system and breast disorders) | 1 (1) | 3 (3)
Vulval disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Scar Pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was limited by poor adherence to the clinical protocol and by incomplete data recovery. Analysis of efficacy-related endpoints was not possible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No